CLINICAL TRIAL: NCT01035268
Title: Adipose Tissue Transfer for Moderate Breast Cancer Conservative Treatment Sequella. Adipocyte Transplant for Esthetical Relapse Treatment of Breast Conservative Treatment
Brief Title: Adipose Tissue Transfer for Moderate Breast Cancer Conservative Treatment Sequella
Acronym: GRATSEC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment rate
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08 SEIN 08
Record Dates: First submitted 2009-12-14; First posted 2009-12-18 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: breast cancer treated by conservative surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- surgery by fatty tissue transfer (Experimental)
  Interventions: Procedure: fatty tissue transfer
- simple supervision (No Intervention)

INTERVENTIONS:
Procedure: fatty tissue transfer — It will be proceeded to aspiration of the fat at the level of the natural steatomeries (hip, stomach), then in a transfer of the fat prepared in the breast by following the standardized protocol.
  Arms: surgery by fatty tissue transfer

SUMMARY:
This is a phase III randomized multi-center study of equivalence comparing the radiological follow-up for patients benefiting from the correction of the esthetical relapse of the preservative treatment by fatty transfer compared with a simple supervision.

It is planned that 440 patients participate in this study which plans to compare 2 groups of patients: a group of patients which will benefit from the surgical treatment by transfer of fatty tissue and a group of patients under simple supervision.

follow-up consultations are planned in 10 in 45 days post-surgery then at 3 months, 6 months, 12 months and 5 years to look for the expected unwanted effects in relation with the surgery but also to estimate the impact of the fatty transfer on the rate of local and\or from a distance relapse.

During these consultations, the surgeon and the patient will also estimate the cosmetic result of the surgery thanks to a questionnaire of cosmetic evaluation and to standardized photos.

ELIGIBILITY:
Inclusion Criteria:

* History of breast cancer treated by conservative surgery .
* Normal inclusion radiological assessment normal (ACR1 or ACR2)
* Moderate Deformations (Type I and II of the classification of Clough).
* Delay with regard to the end of the radiotherapy superior or equal to one-year-old.
* Moderated radio-dystrophies (< Grade 2 of the score LENT/SOMA).
* Signature of the informed consent
* Patient benefiting from social security
* Patient of more than 18 years old

Exclusion Criteria:

* Abnormal radiological assessment (ACR3, ACR4 or ACR5)
* Absence of fatty excess .
* radio surgical relapses with vast fibroses of the breast (> Grade 2 of the score LENT/SOMA).
* Patient under 18 years old.
* administrative difficulties: impossibility to provide enlightened information to the patient, the refusal to sign the consent .
* pregnant women or breast feeding women
* patient under legal guardianship
* bilateral breast cancer regardless histologic type.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2010-02-08 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Verify that the disturbances of the radiological follow-up in 1 year will not be more frequent for the patient benefiting from fatty transfer with regard to a simple surveillance. | 1 year

SECONDARY OUTCOMES:
Estimate the technique on the cosmetic plan : On the quality and on the stability of the result. On the satisfaction of the patient. | 1 year
Estimate the technique on the carcinological plan : Estimate the rate of local relapse and\or in distance. Estimate the rate of survival of the patients. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio GARRIDO, MD, Principal Investigator — Institut Claudius Regaud
Locations (23):
- France (23):
  - CHU de Besançon, Besançon
  - Clinique Saint Antoine, Bois-Guillaume
  - CHU Pellegrin, Bordeaux
  - Institut Bergonie, Bordeaux
  - Pole de Sante de Leonard de Vinci, Chambray-lès-Tours
  - Hopital Henri Mondor, Créteil
  - Centre Hospitalier La Croix Rousse, Lyon
  - Hopital Edouard Herriot, Lyon
  - CHR Marseille Conception, Marseille
  - Institut Paoli Calmettes, Marseille
  - Centre Val d'Aurelle, Montpellier
  - Clinique Brétéché, Nantes
  - INSTITUT CURIE - Site Paris, Paris
  - Hopital Saint Louis, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - INSTITUT CURIE - René Huguenin, Saint-Cloud
  - INSTITUT DE CANCEROLOGIE DE L'OUEST - Centre René Gauducheau, Saint-Herblain
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU Rangueil, Toulouse
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif